CLINICAL TRIAL: NCT06146530
Title: Cerina- Cognitive Behavioural Therapy Based Mobile Application for Managing GAD Symptoms: A Pilot Randomized Controlled Trial
Brief Title: Cerina-A Pilot Randomized Controlled Trial
Acronym: Cerina
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cerina Therapeutics (Industry)
Collaborators: University of Ulster (Other); European Commission (Other)
Responsible Party: Principal Investigator, Ozlem Eylem-van Bergeijk, Post Doctoral Research Associate, Cerina Therapeutics
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: FCPSY-22-084
Record Dates: First submitted 2023-11-19; First posted 2023-11-24 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Treatment Adherence; Generalized Anxiety; Treatment Adherence and Compliance
Keywords: e-health, mhealth, Cognitive Behavior Therapy
MeSH Terms: conditions — Treatment Adherence and Compliance; Generalized Anxiety Disorder | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: The study is a single-blind pilot RCT with two conditions: Treatment (i.e., access to Cerina for 6 weeks) and a waitlist control group (i.e., optional campus-based wellbeing services for 6 weeks)
Who Masked: Investigator
Masking Description: The randomization scheme will be derived using random allocation software by the Cerina technical lead who is not involved in the study. Randomization will take place in blocks of 6, and will take place in a 1:1 ratio. All participants will be informed about the condition they are assigned to. Please see below for the study design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Participants in the treatment arm will have access to Cerina for 6 weeks.
  The intervention (Cerina) consists of 7 sessions of Cognitive Behavioural Threapy (CBT) for the treatment of GAD. Each session contains a range of information and tasks/exercises to help the user understand the condition of GAD, the treatment approach, and how it will apply to them.
  Interventions: Device: Treatment
- Wait-list (Active Comparator): Participants in the waiting-list control condition will have access to the campus-based well-being services offered by the Student Wellbeing team.
  Interventions: Device: Treatment

INTERVENTIONS:
Device: Treatment — The intervention consists of 7 sessions of CBT for the treatment of GAD. Each session contains a range of information and tasks/exercises to help the user understand the condition of GAD, the treatment approach, and how it will be applicable to them. The intervention is based on an evidence-based treatment protocol; hence the sessions will flow from one to the other and the user will complete the sessions in a progressive direction. However, they can repeat a session before going on to the next session. Once all sessions have been completed, the user can go back over any of the sessions. There are anxiety management exercises, which the user can go to whenever they wish. There are also a therapy reflection journal and self-care resources including further anxiety management techniques, resources, and podcasts that the user will have access to whenever they want.
  Other Names: Cerina

SUMMARY:
The goal of this pilot Randomized Controlled Trial is twofold: 1) To learn about the feasibility and usefulness of a mobile application for generalised anxiety symptoms (Cerina); 2) To test the preliminary effects of Cerina in reducing generalized anxiety symptoms compared to a waitlist-control group among Ulster University students presenting mild to moderate symptoms of Generalized Anxiety Disorder (GAD) symptoms. The main research questions are:

Is the Cerina app usable and feasible among Ulster University students reporting mild to moderate GAD symptoms? Is there an indication of the effectiveness of the Cerina app in reducing GAD symptoms compared to a wait-list control group among Ulster University students?

* After the baseline assessment, eligible and consenting participants will be randomized to either intervention or to the wait-list control group.
* Those who are allocated to the intervention group will have access to the Cerina app for 6 weeks.
* Those who are in the wait-list control group will wait for 6 weeks until the intervention group finishes the intervention for their access.
* The wait-list control group will have access to the services offered by the Ulster University Student Wellbeing team.
* Participants in both groups will do mid- (at week 3 after their randomization) and post-assessment (At week 6 after their randomization).
* All participants will also be invited to the post-assessment feedback interviews once they complete their post-assessments. The purpose is to have more in-depth information on their views of the Cerina app, the User Interface, the clinical content, the potential facilitators, and barriers to using it in daily life.

DETAILED DESCRIPTION:
The study is a pilot Randomised Controlled Trial (RCT) with two conditions: Treatment and a waitlist control group. Included eligible participants who have completed the baseline questionnaire will be randomized either into the treatment group in which they have access to the Cerina application for six weeks or into the wait-list control group in which they have access to the campus-based wellbeing services (i.e. routine care) until the intervention group completes Cerina. They will then receive access to Cerina. The randomization scheme will be derived using random allocation software by the Cerina technical lead who is not involved in the study.

All participants will be asked to fill in online self-report measures of anxiety, worrying, depression, and general functioning at baseline (t0), at 3 weeks (t1), and 6 weeks (t2). Additionally, semi-structured interviews will be conducted with the participants in both groups at 6 weeks (t2). The topic guide for the interview was developed by the Cerina team based on the Consolidated Framework for Implementation Research (CFIR), and it is finalized in consultation with the Principal Investigator (PI). The core topics included participants' overall experience and perceptions on the usability of the user interface of Cerina, existing pathways and barriers to using the app in daily life, the clinical utility of the application, the contexts in which the implementation of the clinical content take place and the processes of intervention delivery. The data collection will last 40 minutes, will be remote (online via the MS teams account of Ulster University), and will be facilitated by the PI and the researchers from the Ulster University. Sample size will be determined by data saturation, and sampling will be iterative to ensure theoretical saturation.

Intervention The intervention consists of 7 sessions of CBT for the treatment of anxiety and worry symptoms as part of GAD. Each session contains a range of information and tasks/exercises to help the user understand the condition of GAD, the treatment approach, and how it will apply to them. Once all sessions have been completed, the user can go back over any of the sessions. There are anxiety management exercises, which the user can go to whenever they wish. There are also a therapy reflection journal and self-care resources including further anxiety management techniques, resources, and podcasts that the user will have access to whenever they want. The names of the sessions are: Learning about GAD, dealing with worry, managing worry and anxiety, beliefs about worry, managing uncertainty, testing beliefs, review, and therapy blueprint.

Wait-list Control Condition Participants in the waiting-list control condition will have access to the campus-based well-being services offered by the Student Wellbeing team. The Wellbeing team is based on Belfast, Coleraine, and Magee campuses and provides free and confidential support and guidance to students with a broad range of issues, concerns, and challenges, to help them successfully engage in their studies. Student Wellbeing Assistants provide an initial assessment to determine a student's primary need and then Wellbeing Advisers, Student Mental Health Advisers, and Accessibility Advisers are available to provide a variety of solution-focused interventions based on that need. The Accessibility Advisers also help students with disabilities including diagnosed mental health conditions to get additional support and access funded disability support through Disabled Students' Allowance. Each campus team is led by an experienced Student Wellbeing Manager to support the advisers in the management of risk and lead to an efficient and robust response if a Clinical Incident occurs. Additionally, therapeutic counselling support is also available free to students through the external counselling provider via a dedicated 24/7 counselling helpline. The Student Wellbeing Team works closely with the counselling provider to monitor student engagement and promote the service as appropriate.

b. Statistical techniques

Sample size We seek to recruit 90 participants (N=45 in treatment, N=45 in Wait-list control) in total. The audit of the sample sizes for the pilot and feasibility RCTs indicated that the median sample size per arm across all the types of studies was 30 (Bilingham, Whitehead & Julious, 2013). Browne also recommended that 30 participants per condition are needed to estimate a parameter (Browne, 1995). We take a possible dropout rate into account and aim to include 50% more participants than initially required in both conditions.

Outcome measures:

The outcome measures are online (Qualtrics) self-report questionnaires. The primary outcome measure is anxiety symptoms measured by the Generalised Anxiety Disorder Scale-7 (GAD-7). The secondary outcome measures are: worrying measured by the Penn State Worry Questionnaire (PSWQ-PW), depression measured by the Patient Health Questionnaire (PHQ-9), general functioning measured by the Work and Social Adjustment Scale (WSAS), and usability of the intervention measured by the System Usability Scale (SUS) and semi-structured interviews.

Data analysis plan:

The recruitment and consent rates will be carefully monitored according to the CONSORT guidelines. The group allocation procedure will be monitored by the technical lead of Cerina (independent researcher). The response rates to the study questionnaires and the adherence rates will be monitored by Dr. Özlem Eylem-van Bergeijk.

Participants' views on the quality and usability of the User-Interface Design will be investigated through the SUS questionnaire and semi-structured interviews. These interviews will be audio-recorded and transcribed. The transcripts will be analyzed thematically and independently by two researchers in NVivo software.

The preliminary effects of Cerina in reducing elevated levels of anxiety and worry among students will be tested through the linear mixed models in RStudio version 3.6.1. We will compare reductions in primary/secondary outcomes between and within groups across two time points in the intention-to-treat sample, we will use linear mixed models in RStudio version 3.6.1. This method allows the number of observations to vary between participants and handles missing outcome data. The mixed model uses a longitudinal data structure that includes both fixed and random effects. Time (categorical), group (treatment v. wait-list control), and interactions between group and time will be included as fixed effects in mixed models together with a random intercept and random time effect. Differences in least-squares mean (intervention effects) at each time point with 95% confidence intervals will be derived. Cohen's d for the effect of the intervention will be estimated by calculating the difference between estimated means (corrected for baseline) divided by raw pooled standard deviation. A two-sided p < 0.05 indicates statistical significance. Missing data will be handled through multiple imputations.

We will also monitor people's help-seeking behavior throughout the study, and we will look at the differences between those who used Cerina alone compared to those who used Student Wellbeing and/or counselling services in addition to Cerina.

The reliable change index will also be used to evaluate whether participants have reliable and clinically significant change scores from baseline to post-assessment.

ELIGIBILITY:
Inclusion Criteria:

* Having mild to severe self-reported anxiety symptoms. Those who score between 5 and 19 on the GAD7 questionnaire will be accepted as eligible, ,
* 18 years of age and older
* Enrolled as a student at Ulster University (i.e. having a student id number)
* Fluency in English
* Provision of an informed consent
* Having a smartphone (i.e. Android device or iPhone).
* Having an internet connection

Exclusion Criteria:

* Having minimal anxiety symptoms as defined by a score of 5 and below on the GAD7 questionnaire
* Scoring 19 and above on the GAD7 questionnaire
* Having self-reported suicidal thoughts based on their scores on the Patient Health Questionnaire-9 (PHQ9).
* Having recently (within the last 6 weeks) started taking psychotropic medication.
* Not consenting that their contact details (name, surname, email address) will be shared with the Student Wellbeing team (see the safety section)
* Receiving psychological treatment is not part of the exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-04-24 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
The Generalised Anxiety Disorder Scale-7 (GAD-7) | baseline, week 3 and week 6
  GAD-7 is a 7-item self-report scale that identifies and measures the severity of GAD. Scores range from 0 to 21, with a cut-off score of 5 distinguishing between clinical and non-clinical populations. The scale has good psychometric properties

SECONDARY OUTCOMES:
The Penn State Worry Questionnaire (PSWQ-PW) | baseline, week 3 and week 6
  PSWQ-PW is a 15-item inventory assessing both the weekly status of pathological worry and treatment-related changes of worry during the treatment (Stöbber & Bittencourt, 1998). Each item is scored on a 7-point rating scale, ranging from never 0 (never) to 6 (almost always). The total score ranges from 0 to 90 with a high score indicating more worrying. PSWQ-PW shows good reliability and convergent validity
The Patient Health Questionnaire (PHQ-9) | baseline, week 3 and week 6
  PHQ-9 is a 9-item self-report scale that measures depression symptoms. Scores range from 0 to 27, with a score of 10 and above considered to be a clinically significant level of depression. The PHQ-9 has good reliability and validity
The Work and Social Adjustment Scale (WSAS) | baseline, week 3 and week 6
  WSAS is a 5 item self-report measure that assesses functional impairment. Scores range from 0 to 40. The scale assesses the impact on work, home, social and private activities, and personal and family relationships. A score 20 and above is considered to indicate severe functional impairment, scores between 10 and 20 suggest severe but functional impairment, and scores of 10 and less are considered subclinical. The scale has good reliability and validity
Usability | week 3 and week 6
  The System Usability Scale (SUS) is composed of 10 statements that are scored on a 5-point scale of the extent of agreement (score 0 to 100). The reliability is good (Cronbach's alpha 0.91). Interventions with scores of 70 and above are accepted as highly usable (Bangor et al., 2008) and scores between 50 and 70 indicate acceptable usability of an intervention. Interventions with scores of 50 and below are subject to concerns about their usability by the target population and should be investigated further. Additionally, semi-structured interviews will be conducted with the users to have more in-depth understanding of the usability of the Cerina app in real life.

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Leavey, Prof. dr, Principal Investigator — Ulster University
Locations (1):
- Ulster University, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data including self-reported questionnaires completed by the participants at week 3 and week 6 could be shared with other researchers who inquire the research team about an IPD meta-analysis. If this is the case, in line with the Ulster University GDPR, only anonymized data will be shared in a format which is compatible with R and/or excel for the data analysis.
Supporting Information: Analytic Code
Time Frame: The data will be available upon completion of the study (by the end of August 2024) for 10 years.
Access Criteria: The anonymized data will only be available for IPD meta-analyses

REFERENCES:
- [Derived] Eylem-van Bergeijk O, Robinson T, Manktelow M, Olympios M, Poulter S, Mane P, Panagioti M, Condell J, Leavey G. Cerina-Cognitive Behavioral Therapy-Based Mobile App for Managing Generalized Anxiety Disorder Symptoms Among University Students: Results From a Pilot Feasibility Randomized Controlled Trial. JMIR Mhealth Uhealth. 2025 Oct 9;13:e70691. doi: 10.2196/70691. PMID 41066166
- [Derived] Eylem-van Bergeijk O, Poulter S, Ashcroft K, Robinson T, Mane P, Islam M, Condell J, Leavey G. Cerina: cognitive-behavioural therapy-based mobile application for managing GAD symptoms among Ulster University Students in Northern Ireland - a protocol for a pilot feasibility randomised controlled trial. BMJ Open. 2024 Jul 1;14(6):e083554. doi: 10.1136/bmjopen-2023-083554. PMID 38950994
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30211576/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/32950939/